CLINICAL TRIAL: NCT01063270
Title: Randomized Control Trial Comparing Efficacy of Antibiotic Therapy Alone Versus Antibiotic Therapy in Conjunction With Quadruple Pulse Therapy Using NdYag Laser in Treatment of Hidradenitis Suppurativa
Brief Title: Trial Comparing Efficacy of Treatments for Hidradenitis Suppurativa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB5974
Record Dates: First submitted 2010-02-02; First posted 2010-02-05 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Antibiotics; Laser
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Clindamycin; Rifampin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Antibiotics (Active Comparator)
  Interventions: Drug: Clindamycin & Rifampin
- Topical Antibiotics and Laser treatment (Active Comparator)
  Interventions: Procedure: Clindamycin + Rifampin along with NdYag Laser treatment

INTERVENTIONS:
Drug: Clindamycin & Rifampin — Clindamycin 300mg twice daily for 10 weeks and Rifampin 300mg twice daily for 10 weeks
  Arms: Oral Antibiotics
Procedure: Clindamycin + Rifampin along with NdYag Laser treatment — Clindamycin 300mg twice daily for 2 weeks Rifampin 300mg twice daily for 2 weeks along with 3 NdYag laser sessions.
  Arms: Topical Antibiotics and Laser treatment

SUMMARY:
The purpose of this research study is to further evaluate the efficacy of two treatment regimens for the treatment of hidradenitis suppurativa. This is a randomized controlled study. Patients will be randomly assigned to an arm of the study.

DETAILED DESCRIPTION:
Histological studies suggest that HS is a disease of the follicles with apocrine involvement as a secondary event. The investigators have identified in a previous study that the Nd Yag laser is highly effective for decreasing the inflammation, pain, suppuration and frequency of recurrence of HS. Oral antibiotic therapy with Clindamycin and Rifampin has also been reported in previous studies to be a highly effective treatment regimen for HS and is commonly used by physicians in medical management of HS. The investigators would like to compare the efficacy of NdYag laser treatment combined with antibiotics versus treatment with antibiotics alone. The goal is to evaluate the success of these two treatment regimens on existent HS lesions as well as prevention of recurrence. There will be approximately 18 people in this research study at Henry Ford Health System (HFHS).

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 16 years old and weigh a minimum of 80lbs. Weight requirement is for the purpose of maintaining safe clindamycin and rifampin dosing regimens.
2. Be otherwise healthy
3. Have a diagnosis of HS
4. Patients must have Hurley stage II HS, with one or more widely separated recurrent abscesses, with tract and scarring. Involvement should be bilateral and symmetric on axillae, inguinal regions or inframammary regions
5. Agree to abide by the Investigator's guidelines regarding photosensitizing drugs
6. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form
7. Agree to follow and undergo all study-related procedures

Exclusion Criteria:

1. Patients with HS Hurley stage I and III will be excluded from participation in the study
2. Patients who are currently pregnant will not be able to take part in the study due to the unknown effects of antibiotics
3. Concomitant use of systemic or topical treatments for HS not involved in current study. Patients must discontinue all forms of oral therapy as systemic and topical antibiotics and retinoids for 2 weeks prior to the start of any treatment
4. Exacerbation of the patient's original condition expressed clinically by a shift from Hurley Stage II to Stage III
5. Patient is unable to take antibiotic therapy
6. Any reason the investigator feels the patient should not participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-02; Primary Completion 2011-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number and severity of lesions | 5 total clinic visits over 6 month period

SECONDARY OUTCOMES:
Change in quality of life during treatment | 5 total clinic visits over 6 month period
Recurrence of disease | 5 total clinic visits over 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat Hamzavi, M.D., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital Department of Dermatology. 3031 West Grand Blvd, Suite 800, Detroit, Michigan, United States